CLINICAL TRIAL: NCT00186420
Title: Adjuvant Taxotere in Patients With High Risk Prostate Cancer Post Prostatectomy and Radiation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sandy Srinivas, Associate Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PROS0004
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Taxotere
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Taxotere

SUMMARY:
The purpose of this study is to evaluate time to progression (TTP) by PSA in patients with high risk prostate cancer after definitive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a radical prostatectomy (should have unmeasurable PSA) or radiation therapy for prostate cancer and who have high risk disease as defined by one of the following:

  * Node positive disease post-operatively
  * Capsule involvement
  * Seminal Vesicles involvement
  * Gleason score ≥ 8
  * >50% of core biopsies that are positive
  * Clinical Stage T2c and T3
  * Pre-op PSA > 15 plus Gleason score of 7

    * Age greater than 18
    * ECOG Performance Status 0-1
    * Serum creatinine <= 1.5 mg/dl
    * Granulocyte count >= 1500/m3, Hemoglobin > 8.0 g/dl, and platelet count >= 100,000/m3
    * Total bilirubin <= ULN
    * AST, ALT and Alkaline Phosphatase must be within the range allowing for eligibility.
    * Signed patient informed consent.
    * Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for three months thereafter.

Exclusion Criteria:

* Peripheral neuropathy > grade 1
* History of severe hypersensitivity to Taxotere® or other drugs formulated with polysorbate 80.
* Patients who have received previous chemotherapy or are being treated on another clinical trial using an investigational agent.
* Active infection within 14 days of beginning treatment
* Patients with a serious illness or medical condition, history of significant neurologic or psychiatric or active infection.
* Patients with a current malignancy. Patients with prior a history of in situ lobular carcinoma of the breast, basal or squamous cell skin cancer, are eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-07; Primary Completion 2006-01 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To evaluate time to progression (TTP) by PSA in patients with high risk prostate cancer after definitive therapy. | Following treatment

SECONDARY OUTCOMES:
To evaluate the toxicity of taxotere and hormones given adjuvantly. | Following treatment
To measure Quality of Life on this therapy. | Following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Srinivas, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Center, Stanford, California, United States